CLINICAL TRIAL: NCT00738972
Title: Left Ventricular Hypertrophy Reduction With Statins in Hypertensives Patients.
Brief Title: Left Ventricular Hypertrophy Reduction With Statins in Hypertensives Patients (MK0653A-168)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated early due to sample size, not possible to perform further statistical analysis.
Sponsor: Fundación Lindavista del Corazón AC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MK-0653A-168; 2008_020; NCT00621127 (obsolete NCT alias)
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Results first posted 2013-08-13 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Pravastatin; Simvastatin; Ezetimibe, Simvastatin Drug Combination

ARMS (4):
- Valsartan 80 mg + Paravastin 40 mg (Active Comparator): Participants who were administered Valsartan 80 mg plus paravastin 40 mg by mouth daily for one year. (Group A)
  Interventions: Drug: valsartan; Drug: pravastatin
- Valsartan 80 mg + Simvastatin 40 mg (Active Comparator): Participants who were administered Valsartan 80 mg plus simvastatin 40 mg by mouth daily for one year. (Group B)
  Interventions: Drug: valsartan; Drug: simvastatin
- Valsartan 80 mg + Simvastatin 40 mg / Ezetimibe 10 mg (Experimental): Participants who were administered Valsartan 80 mg plus simvastatin 40 mg / ezetimibe 10 mg by mouth daily for one year. (Group C)
  Interventions: Drug: valsartan; Drug: ezetimibe (+) simvastatin
- Valsartan 80 mg (Active Comparator): Participants who were administered Valsartan 80 mg by mouth daily for one year. (Group D)
  Interventions: Drug: valsartan

INTERVENTIONS:
Drug: valsartan — 80 mg valsartan. Duration: 12 months. Tablets
  Other Names: Diovan
Drug: pravastatin — 40 mg pravastatin. Duration: 12 months. Tablets
  Other Names: Pravacol
  Arms: Valsartan 80 mg + Paravastin 40 mg
Drug: simvastatin — 40 mg simvastatin. Duration: 12 months. Tablets
  Other Names: Zocor; MK0733
  Arms: Valsartan 80 mg + Simvastatin 40 mg
Drug: ezetimibe (+) simvastatin — ezetimibe (+) simvastatin 10/40 mg. Duration: 12 months. Tablets
  Other Names: vytorin; MK0653A
  Arms: Valsartan 80 mg + Simvastatin 40 mg / Ezetimibe 10 mg

SUMMARY:
Evaluate pleiotropic effects of simvastatin in hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Females Or Males Over 18 Years Old
* Patients With Systemic Arterial Hypertension Grade I And II According With The European Society Of Cardiology
* Left Ventricular hypertrophy Demonstrated By Echocardiography
* Mild To Moderated hypercholesterolemia
* Willing To Participate And Sign The Informed Consent Form (ICF)

Exclusion Criteria:

* Type 1 Or 2 Diabetes Mellitus
* Familiar hypercholesterolemia
* Low Density Lipoprotein-Cholesterol (LDL-C) > 190 mg/dl
* History Of Myocardial Infarction Or Stable Chronic Angina
* Triglycerides >250 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valsartan 80 mg + Paravastin 40 mg | Valsartan 80 mg + Simvastatin 40 mg | Valsartan 80 mg + Simvastatin 40 mg / Ezetimibe 10 mg | Valsartan 80 mg
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan 80 mg + Paravastin 40 mg | Valsartan 80 mg + Simvastatin 40 mg | Valsartan 80 mg + Simvastatin 40 mg / Ezetimibe 10 mg | Valsartan 80 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 11
Age, Customized [Number; unit: participants]
  >18 years | 3 | 3 | 3 | 2 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 8
  Male | 1 | 1 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Hypertrophy Reduction With Statins in Hypertensive Patients
Description: Left ventricular hypertrophy reduction was to be measured by echocardiography.
Time Frame: 6 Month(s)
Population: This study was terminated early and due to sample size it was not possible to perform further statistical analyses.
Arm/Group | Valsartan 80 mg + Paravastin 40 mg | Valsartan 80 mg + Simvastatin 40 mg | Valsartan 80 mg + Simvastatin 40 mg / Ezetimibe 10 mg | Valsartan 80 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Valsartan 80 mg + Paravastin 40 mg | Valsartan 80 mg + Simvastatin 40 mg | Valsartan 80 mg + Simvastatin 40 mg / Ezetimibe 10 mg | Valsartan 80 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/2

LIMITATIONS AND CAVEATS:
This study was terminated early and due to sample size it was not possible to perform further statistical analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No